CLINICAL TRIAL: NCT01737866
Title: An Open-label, Single-dose Study of the Safety, Tolerability, and Pharmacokinetics of AMG 423 in Healthy Subjects and Subjects With Various Degrees of Renal Insufficiency and Effect of Hemodialysis on AMG 423 Pharmacokinetics
Brief Title: Pharmacokinetics Study of AMG 423 in Healthy Subjects and Subjects With Various Degrees of Renal Insufficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080676
Record Dates: First submitted 2012-10-16; First posted 2012-11-30 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure
Keywords: Heart, Failure, Renal, Insufficiency, Cardiac, Kidney, Hemodialysis, Impairment, omecamtiv mecarbil, cardiac myosin activator, CK-1827452
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): End Stage Renal Diseas (ESRD) requiring hemodialysis
  Interventions: Drug: AMG 423
- Group 2 (Experimental): Normal renal function (eGFR >or = 80mL/min/1.73m^2)
  Interventions: Drug: AMG 423
- Group 3 (Experimental): Mild decrease in GFR (eGFR 60-79 mL/min/1.73m^2)
  Interventions: Drug: AMG 423
- Group 4 (Experimental): Moderate decrease in GFR (eGFR 30-59 mL/min/1.73m^2)
  Interventions: Drug: AMG 423
- Group 5 (Experimental): Severe decrease in GFR (eGFR 15-29 mL/min/1.73m^2)
  Interventions: Drug: AMG 423
- Group 6 (Experimental): Normal renal function (eGFR >or = 80mL/min/1.73m^2)
  Interventions: Drug: AMG 423

INTERVENTIONS:
Drug: AMG 423 — omecamtiv mecarbil

SUMMARY:
A phase 1, open-label study in subjects with normal renal function and subjects with various degrees of renal insufficiency, including patients with end-stage renal disease (ESRD) requiring hemodialysis. The primary objective is to evaluate the single-dose PK of AMG 423 in subjects with various degrees of renal insufficiency, including patients with end-stage renal disease requiring hemodialysis.

DETAILED DESCRIPTION:
This study was conducted by Amgen as the IND holder, with Cytokinetics as a collaborator. Due to the termination of the collaboration agreement between Amgen and Cytokinetics in May 2021 and subsequent transfer of the omecamtiv mecarbil IND from Amgen to Cytokinetics, Cytokinetics is now listed as the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years of age
* Laboratory test values (clinical chemistry and hematology)within normal limits, (other than test values out of the normal range for subjects with CKD [groups 1 and 3 through 5]), or clinically acceptable to the investigator and sponsor at screening and day -3
* Free of any clinically significant disease or condition(s) (other than that consistent with CKD for subjects in groups 1 and 3 through 5) that require a physician's care and/or would interfere with the evaluations, procedures, or participation in the study per the investigator's discretion;

Exclusion Criteria:

* Subjects whose second MDRD eGFR result during the screening period is not within 10% of the first eGFR result
* Subjects who have received a functioning renal transplant within the past year
* Subjects with ESRD who do not have a functioning hemodialysis access
* Subjects with hemodynamic instability during hemodialysis
* Subjects whose renal insufficiency is due to active autoimmune renal disease
* Subjects with renal insufficiency or ESRD requiring hemodialysis and Troponin I > upper limit of normal (ULN) at screening or day -3
* Subjects with history of heart disease or unstable angina within the last 3 months
* Subjects with uncontrolled diabetes (Hb1Ac > 8%) and/or subjects who are able but unwilling to adhere to the required fasting intervals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
AMG 423 Pharmacokinetic Parameters | Twenty time points, up to eight days
  Part A and Part B: Total AMG 423 pharmacokinetic parameters including area under the plasma concentration time curve (AUC) from time 0 to the time of the last quantifiable sample (AUC0-t) and maximum observed plasma concentration after dosing (Cmax).

SECONDARY OUTCOMES:
Other Total AMG 423 PK Parameters | Twenty time points, up to eight days
  Total AMG 423 pharmacokinetic parameters including but not limited to terminal phase half life (t1/2) and time of maximum AMG 423 plasma concentration (tmax), AUC from time 0 to infinity (AUCinf) and apparent plasma clearance (CL/F) for Part A and Part B;
AMG 423 Dialysis Clearance | Hours 4, 5, 6, 7 & 8 post-dose
  AMG 423 dialysis clearance (CLd) for ESRD subjects in Part A;
AMG 423 Metabolites | Twenty time points, up to eight days
  AMG 423 metabolites (M3 and M4) pharmacokinetic parameters including but not limited to AUC0-t, AUCinf, AUC metabolite to parent ratios, Cmax, tmax and t1/2, if appropriate.
Safety | Up to 46 days, including a 28 day screening period
  Secondary safety endpoints are subject incidence of adverse events and clinically significant changes in vital signs, physical examinations, clinical laboratory tests and ECGs.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Orlando, Florida, United States

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com